CLINICAL TRIAL: NCT02938338
Title: Physical Activity, Sedentary and Energy Consumption After Bariatric Surgery
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Region Örebro County (Other)
Responsible Party: Principal Investigator, Lars Hagberg, PhD, Region Örebro County
Other Study IDs: Regionorebrolan 001
Record Dates: First submitted 2015-04-28; First posted 2016-10-19 (Estimated); Last update posted 2016-10-19 (Estimated); Status verified 2016-10

CONDITIONS: Sedentary Lifestyle
MeSH Terms: conditions — Sedentary Behavior | interventions — Bariatric Surgery

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Obese patients with BMI above 35: Bariatric surgery
  Interventions: Procedure: Bariatric surgery

INTERVENTIONS:
Procedure: Bariatric surgery — Bariatric surgery, with an anticipated mean weight loss of 30 kg

SUMMARY:
The aim is

to examine the energy consumption before and after bariatric surgery. The study will contribute to the knowledge if operations should be complemented by interventions to increase energy expenditure, mainly by reducing sedentary.

as input for the design of an intervention to reduce sedentary. Such intervention should be based on knowledge of the mediators of physical activity among the subjects that need to be strengthened.

DETAILED DESCRIPTION:
The aim is

to examine the energy consumption before and after bariatric surgery. The study will contribute to the knowledge if operations should be complemented by interventions to increase energy expenditure, mainly by reducing sedentary.

as input for the design of an intervention to reduce sedentary. Such intervention should be based on knowledge of the mediators of physical activity among the subjects that need to be strengthened.

Hypothesis Patients who undergo bariatric surgery have before surgery low energy consumption related to physical activity. The investigators hypothesis is that low energy consumption for the most part retained and that is independent of whether one starts exercising or not.

About the level of physical activity and energy expenditure Increased physical activity after obesitasoperation is correlated with greater weight loss. According the Swedish Obesitas Surgery study, the percentage of persons who were classified as physically inactive decreased from 45% before surgery to less than 10% 6 months after surgery. The proportion of inactive people 6 years after surgery was 20%. Patients who undergo surgery for obesity has low energy consumption related to physical activity before surgery, as measured by pedometer or self-reported physical activity. The results in terms of increased physical activity after surgery are contradictory, where physical activity increases more in studies based on self-reported physical activity than in studies where measurements are made with the objective method. In a Swedish study (n = 56 women) no change could be seen in physical activity and sedentary after bariatric surgery. For a group of extremely obese (BMI around 50) were found reduced energy consumption by 25% after surgery. The decrease was related to lower body weight (average 53 kg) and thus decreased basal energy consumption and lower energy consumption during physical activity. A 20% decrease in body weight means an average of 400 kcal / day lower energy consumption.

Among adults is the basal energy consumption approximately 1,500 kcal per day (depending on body size). For adults, the average energy consumption related to physical activity 300 kcal / day, compared with 1000 kcal / day for people who traditionally live (hunter / gatherers). Patients who undergo bariatric surgery have weak mediating factors for physical activity.

About sedentary Sedentary and low energy consumption is a risk factor for cardiovascular disease, type 2 diabetes and premature death, even after correction for exercise / training and body mass index (BMI). Sedentary is also a contributing factor to obesity, independent of physical activity in general. Moving in everyday life (apart from exercise) is an essential part of the investigators energy consumption. The difference in energy consumption between a mainly sedentary person and a person who has a relatively moving life, may be 700 kcal per day) and compared with a very physically active (moving much at work and leisure), the difference be 2000 kcal per day. Among people with overweight or obesity, moving in everyday life is responsible for 90% of the energy consumption related to physical activity. Overweight people are sedentary 2-2.5 hours more per day than normal weight people, and that corresponding to a difference in energy of 350 kcal / day. In one year, that is equivalent to 15 kg of body weight. For the population as a whole, 60% of waking hours is sedentary.

About behavioral change and interventions to reduce sedentary For patients undergoing bariatric surgery are increased physical activity in everyday life / decreased sedentary very important for a positive weight development and favorable results regarding the health and quality of life, but low energy consumption in everyday life may remain after surgery.

It is difficult to change an established behavior, or a habit, well documented in social cognitive theory. Within this theoretical framework has also behavioral change models been developed. According to Nilsen et al is a habit behavior that has been repeated until it has become more or less automatically and is independently of the active awareness of what is happening. Gradually changing behavior control from being guided by beliefs, attitudes and intentions, that is triggered by a particular situation or context. It has been shown that behaviors that are repeated in a constant, unchanged context are difficult to change. So, change in the context where the habit has been established should to be important for a successful change of a habitual behavior.

Generally, there is lack of efficacy studies of interventions to reduce sedentary. A meta-analysis of interventions to reduce sedentary among adolescents show a small but significant effect. The focus in interventions and research should be on decreased sedentary connected to television and computer use, sitting at workplace and sitting in the car.

About mediating factors for increased physical activity and decreased sedentary Mediating factors for increased physical activity are factors that pave the way for change to come about and continue. The best evidence available for self-efficacy (situation-bound self-confidence, for example, "I know that I can take uo training again after a break."), social support (support and encouragement from family and friends) and enjoyment (experience / joy of movement).

ELIGIBILITY:
Inclusion Criteria:

* All patient at Lindesbergs hospital that get bariatric surgery (a limit to get the surgery is BMI above 35)

Exclusion Criteria:

* Not understanding Swedish or English
* Not the first bariatric surgery

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients undergoing bariatric surgery
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2015-06; Primary Completion 2018-12 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Calories consumed | One year after surgery
  Amount calories consumed per day
Hours sedentary | One year after surgery
  Hours sedentary during a day

SECONDARY OUTCOMES:
Mediators of physical activity | One year after surgery
  Self-efficacy, social support and enjoyment of physical activity measured by questionaires

CONTACTS AND LOCATIONS:
Overall Officials: Lars A Hagberg, PhD, Principal Investigator — Region Örebro County
Locations (1):
- Region Örebro län, Örebro, Örebro County, Sweden

IPD SHARING:
Plan to Share IPD: Undecided